CLINICAL TRIAL: NCT01158742
Title: Live Kidney Donor Study -Renal Function Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE-06
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Kidney Donation; Kidney Failure; Kidney Transplantation
Keywords: Glomerular Filtration Rate
MeSH Terms: conditions — Renal Insufficiency | interventions — Glomerular Filtration Rate; Iothalamic Acid; Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Caucasians who donated a kidney at Mayo Clinic in Rochester, Minnesota (MN)
  Interventions: Other: Glomerular Filtration Rate with Iothalamate
- 2: Caucasians who donated a kidney at the University of Minnesota
  Interventions: Other: Glomerular Filtration Rate with Iohexol
- 3: African-Americans who donated a kidney at the University of Alabama
  Interventions: Other: Glomerular Filtration Rate with Iothalamate

INTERVENTIONS:
Other: Glomerular Filtration Rate with Iothalamate — used to determine kidney function
  Other Names: GFR
  Groups: 1; 3
Other: Glomerular Filtration Rate with Iohexol — used to determine kidney function
  Other Names: GFR
  Groups: 2

SUMMARY:
Kidney transplantation from living donors has been shown to carry many benefits over deceased donor transplantation. Because of benefits such as shorter waiting times and improved outcome for transplant recipients, living kidney donation accounts for an increasing number of kidney transplants nationwide. Most published studies about living kidney donation demonstrate that the procedure is safe, but they also emphasize concerns that long-term data on live donor outcomes are insufficient. In particular, data concerning the extent of renal function decline after donation are inadequate. This study will measure glomerular filtration rate (GFR) in previous living donors and aims to more accurately describe renal function after kidney donation.

DETAILED DESCRIPTION:
Previous studies poorly describe renal function after kidney donation. Most published studies of renal function after donation are based on predictive equations, which were not designed for living kidney donors. One concern is that use of these equations may underestimate glomerular filtration rate (GFR) following donation. Systematic underestimation of GFR may cause previous kidney donors to be inaccurately categorized as having chronic kidney disease (CKD).

While data for the entire kidney donor population are insufficient, there is even less available information about renal function after donation in black renal donors. In the general population, the incidence of end stage renal disease is higher among blacks compared to whites. Whether this pattern carries over to the black renal donor population is unclear.

The primary objectives of this study are to more accurately measure current GFR; evaluate the change in GFR before and after donation; compare measured GFR in donors matched by race, age, sex, time from donation, presence of hypertension, and presence of obesity; and evaluate differences between predictive equations and measured GFR.

This is an observational study to look at the long term outcomes in living kidney donors. Participants in this study will also be participants in DAIT RELIVE-04. As a part of this study, participants will have a brief medical history taken and a glomerular filtration rate test performed.

ELIGIBILITY:
Inclusion Criteria:

* Underwent unilateral donor nephrectomy between 5 and 50 years ago; but no later than June 30, 2005 at Mayo Clinic or University of Minnesota
* Alive at the time of study recruitment
* Underwent GFR measurement before and early after donor nephrectomy (Mayo Clinic participants only)
* Underwent GFR measurement late after donor nephrectomy and 3 or more years prior to the invitation to participate in this study (UMN participants only)
* Self reported black race (UAB participants only)
* Negative serum pregnancy test (Total Beta Human Chorionic Gonadotropin (HCG) <5) for women of child-bearing potential

Exclusion Criteria:

* Less than 5 years out from time of kidney donation
* Inability to contact donor
* Inability or unwillingness to provide informed consent
* Iodine or iodinated contrast allergy.
* Pregnant or breast feeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals participating in DAIT RELIVE-04 who donated a kidney at the Mayo Clinic-Rochester, University of Minnesota, or the University of Alabama
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in measured GFR from before donor nephrectomy compared to early (within first 2 years) after donor nephrectomy. | Throughout study
Change in measured GFR from early after donor nephrectomy compared to late donor nephrectomy. Change in measured GFR from early to late after donor nephrectomy stratified by: time since donation, hypertensive donors, obese donors, and age of donors | Throughout study
Differences in measured GFR in black donors compared to white donors matched by age, sex and time from donation | Throughout study
Incremental differences between measured GFR and estimated GFR before donor nephrectomy, early after donor nephrectomy, and late after donor nephrectomy | Throughout study

SECONDARY OUTCOMES:
Differences in measured GFR between hypertensive donors and normotensive donors | Throughout study
Differences in measured GFR between donors with familial history of renal disease (LRD) and donors without familial history of renal disease (LURD) | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Taler, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Taler SJ, Messersmith EE, Leichtman AB, Gillespie BW, Kew CE, Stegall MD, Merion RM, Matas AJ, Ibrahim HN; RELIVE Study Group. Demographic, metabolic, and blood pressure characteristics of living kidney donors spanning five decades. Am J Transplant. 2013 Feb;13(2):390-8. doi: 10.1111/j.1600-6143.2012.04321.x. Epub 2012 Nov 8. PMID 23137211
- [Result] Jacobs CL, Gross CR, Messersmith EE, Hong BA, Gillespie BW, Hill-Callahan P, Taler SJ, Jowsey SG, Beebe TJ, Matas AJ, Odim J, Ibrahim HN; RELIVE Study Group. Emotional and Financial Experiences of Kidney Donors over the Past 50 Years: The RELIVE Study. Clin J Am Soc Nephrol. 2015 Dec 7;10(12):2221-31. doi: 10.2215/CJN.07120714. Epub 2015 Oct 13. PMID 26463883
- [Result] Jowsey SG, Jacobs C, Gross CR, Hong BA, Messersmith EE, Gillespie BW, Beebe TJ, Kew C, Matas A, Yusen RD, Hill-Callahan M, Odim J, Taler SJ; RELIVE Study Group. Emotional well-being of living kidney donors: findings from the RELIVE Study. Am J Transplant. 2014 Nov;14(11):2535-44. doi: 10.1111/ajt.12906. Epub 2014 Oct 7. PMID 25293374
- [Result] Gross CR, Messersmith EE, Hong BA, Jowsey SG, Jacobs C, Gillespie BW, Taler SJ, Matas AJ, Leichtman A, Merion RM, Ibrahim HN; RELIVE Study Group. Health-related quality of life in kidney donors from the last five decades: results from the RELIVE study. Am J Transplant. 2013 Nov;13(11):2924-34. doi: 10.1111/ajt.12434. Epub 2013 Sep 6. PMID 24011252
- [Result] Noppakun K, Cosio FG, Dean PG, Taler SJ, Wauters R, Grande JP. Living donor age and kidney transplant outcomes. Am J Transplant. 2011 Jun;11(6):1279-86. doi: 10.1111/j.1600-6143.2011.03552.x. Epub 2011 May 12. PMID 21564530
- [Result] Messersmith EE, Gross CR, Beil CA, Gillespie BW, Jacobs C, Taler SJ, Merion RM, Jowsey SG, Leichtman AB, Hong BA; RELIVE Study Group. Satisfaction With Life Among Living Kidney Donors: A RELIVE Study of Long-Term Donor Outcomes. Transplantation. 2014 Dec 27;98(12):1294-300. doi: 10.1097/TP.0000000000000360. PMID 25136843
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY291 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY291 — ImmPort study identifier is SDY291
- Available data/document: Study Protocol: SDY291 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY291 — ImmPort study identifier is SDY291. The study protocol is available through the Design tab on the site.
- Available data/document: Study summary, -design, -demographics, -files: SDY291 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY291 — ImmPort study identifier is SDY291